CLINICAL TRIAL: NCT01030185
Title: A Prospective, Multi-center, Open Label, Non-randomized Study to Investigate the Safety and Performance of the Automated Fluid Shunt in Patients With Ascites and Diuretic Resistance
Brief Title: Safety and Performance of the Automated Fluid Shunt in Patients With Ascites and Diuretic Resistance
Acronym: PIONEER
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NovaShunt AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-AAR-002
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Ascites
Keywords: ascites; liver cirrhosis
MeSH Terms: conditions — Ascites; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NovaShunt's Automated Fluid Shunt (Experimental): The Automated Fluid Shunt (AFS) Device
  Interventions: Device: NovaShunt's Automated Fluid Shunt implantation

INTERVENTIONS:
Device: NovaShunt's Automated Fluid Shunt implantation — The Automated Fluid Shunt (AFS) Device consists of an implantable sealed housing which contains an internally powered pump with supportive electronic components and circuits, an implantable Peritoneal Catheter, implantable Bladder Catheter and a non-implantable Charger used for wireless recharging an AFS battery and collecting data from the Device.
  Other Names: NovaShunt

SUMMARY:
To investigate the safety and performance of the Automated Fluid Shunt in patients with ascites and diuretic resistance.

Study Size and Duration The primary study population will include 40 patients enrolled and implanted with the NovaShunt Automated Fluid Shunt (AFS) in up to 15 centers in Europe.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Recurrence of ascites defined as clinical reappearance of ascites within 4 weeks of initial paracentesis.
* Cirrhosis of any etiology
* Failure to respond to a maximum of 160 mg/d of furosemide and 400 mg/d of spironolactone (or equivalent doses of loop-acting and distal-acting diuretics), or intolerance to high dose diuretics because of hyponatremia, hyperkalemia, or other side-effects
* Dietary sodium restriction <88mEq/d.
* Serum creatinine levels of ≤ 2.0 mg/dL for at least 7 days before study entry.
* Total bilirubin levels of less than 3 mg/dL.
* Expected survival of greater than 6 months
* Written informed consent
* Ability to comply with study procedures and ability to operate the device.
* Women of childbearing age should use adequate contraceptives

Exclusion Criteria:

* Presence of recurring systemic or local infection, such as peritonitis, urinary tract infection, or abdominal skin infection.
* Presence of peritoneal carcinomatosis
* Advanced hepatocellular carcinoma, demonstrated by:

  1. One tumor that is >5 cm diameter
  2. 3 or more nodules of >3 cm diameter
  3. Portal thrombosis
* Other evidence of a malignant Etiology for Ascites
* Evidence of extensive ascites loculation
* Gastrointestinal hemorrhage due to portal hypertension in the 2 weeks prior to the inclusion in the study.
* Hepatic encephalopathy in the two weeks prior to implant
* Presence of a TIPS or surgical portosystemic shunt
* Presence of Budd-Chiari syndrome
* Previous liver transplant
* Obstructive uropathy
* Coagulopathy that could not be corrected to a prothrombin time INR <1.8,
* Thrombocytopenia that could not be corrected to a platelet count greater than 60,000/mm3
* Any other clinically significant disease that could be adversely affected by study participation judged by the Investigator
* Any condition requiring emergency treatment
* Pregnancy
* Patients being in another clinical study that did not reach primary endpoint yet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The safety of the NovaShunt AFS will be evaluated by the incidence and severity of device- and procedure-related serious adverse events | 6 months

SECONDARY OUTCOMES:
Paracentesis requirements | 6 month
Hematology | 6 month
Incidence of hemodynamic instability | 6 month
Incidence and severity of peripheral edema | 6 month
Patient Quality of Life. | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Jose Such, MD, Principal Investigator — Hospital General Uneversitario de Alicante C/ Maestro Alonso 109 - 03010 Alicante /Alacant, Spain
Locations (9):
- Department of hepatology, UZ Leuven, campus Gasthuisberg, Leuven, Belgium
- Bulgaria (2):
  - Clinic of Internal Diseases, MHAT "Tokuda Hospital Sofia" JSC, Sofia
  - Military Medical Academy, Clinica of Gastroenterology and Hepatology, Sofia
- Germany (4):
  - Medizinische Klinik mit Schwerpunkt Hepatologie und Gastroenterologie Charité, Campus Virchow Klinikum, Berlin
  - Medizinische Klinik und Poliklinik I, Bonn
  - Klinikum und Fachbereich Medizin Johann Wolfgang Goethe-Universität, Frankfurt
  - Universitätsklinikum Regensburg, Regensburg
- Spain (2):
  - Hospital General Uneversitario de Alicante, Alicante
  - Hospital de la Santa Pau I Sant Creu, Barcelona